CLINICAL TRIAL: NCT07376551
Title: The Effect of Isokinetic Strength on Anaerobic Capacity in Recreationally Active Young Adult Males
Brief Title: Isokinetic Strength and Anaerobic Capacity
Acronym: ISAC
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ramiz ARABACI, Uludağ university, Uludag University
Other Study IDs: E-87914409-050.04-117159
Record Dates: First submitted 2026-01-09; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult; Physical Condition
Keywords: Physical Fitness; Exercise Test; Acute Exercise

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low Anaerobic Power (LAP): Participants are recreationally active young adult males classified into three cohorts based on relative peak power (W/kg) obtained from the Wingate Anaerobic Test. The low, moderate, and high anaerobic power groups represent individuals with differing anaerobic performance capacities derived from median-based classification. All participants are physically active but non-elite, with no recent history of orthopedic injury or cardiopulmonary disease. Comparisons among cohorts are conducted to examine differences in isokinetic knee extensor and flexor strength parameters.
- Moderate Anaerobic Power (MAP): Participants are recreationally active young adult males classified into three cohorts based on relative peak power (W/kg) obtained from the Wingate Anaerobic Test. The low, moderate, and high anaerobic power groups represent individuals with differing anaerobic performance capacities derived from median-based classification. All participants are physically active but non-elite, with no recent history of orthopedic injury or cardiopulmonary disease. Comparisons among cohorts are conducted to examine differences in isokinetic knee extensor and flexor strength parameters.
- High Anaerobic Power (HAP): Participants are recreationally active young adult males classified into three cohorts based on relative peak power (W/kg) obtained from the Wingate Anaerobic Test. The low, moderate, and high anaerobic power groups represent individuals with differing anaerobic performance capacities derived from median-based classification. All participants are physically active but non-elite, with no recent history of orthopedic injury or cardiopulmonary disease. Comparisons among cohorts are conducted to examine differences in isokinetic knee extensor and flexor strength parameters.

SUMMARY:
This study aims to investigate differences in isokinetic knee extensor and flexor strength parameters among recreationally active young adult males classified into low, moderate, and high anaerobic power groups based on relative peak power (W/kg) obtained from the Wingate Anaerobic Test. Eighty male participants aged 22-30 years, engaging in regular physical activity, will undergo body composition analysis, isokinetic strength testing at 60°/s, and a 30-second Wingate test performed on separate days. Participants will be grouped according to median-based anaerobic power classification to allow meaningful group comparisons. Group differences in peak torque and total work will be analyzed using ANOVA or non-parametric equivalents, and relationships between Wingate parameters and isokinetic strength will be examined using correlation analyses. The findings are expected to provide novel insights into the relationship between anaerobic power classification and lower-extremity muscle strength profiles, contributing to performance profiling and training planning in recreationally active populations.

DETAILED DESCRIPTION:
This study will investigate the relationship between anaerobic power classification and isokinetic lower-extremity muscle strength in recreationally active young adult males. Participants will be classified into three anaerobic power groups (low, moderate, and high) based on relative peak power (W/kg) obtained from the Wingate Anaerobic Test. This classification approach is intended to move beyond single-variable correlation analyses commonly reported in the literature and to enable meaningful group-based comparisons of muscle strength profiles.

A total of 80 male participants aged 22-30 years who engage in regular physical activity at least twice per week will be recruited. Individuals with a history of serious orthopedic injury within the past six months, cardiovascular or respiratory disease, or regular medication use will be excluded. Body composition parameters will be assessed using bioelectrical impedance analysis prior to performance testing.

Isokinetic knee extensor and flexor strength of the dominant leg will be evaluated using concentric contractions at an angular velocity of 60°/s. Peak torque and total work values will be recorded as primary isokinetic strength outcomes. Anaerobic performance will be assessed on a separate day using a 30-second Wingate Anaerobic Test performed on a cycle ergometer, during which participants will be verbally encouraged to exert maximal effort throughout the test. Relative peak power, mean power, and fatigue index values will be obtained.

Participants will be grouped according to median-based classification of relative peak power values to facilitate comparison among anaerobic power levels in a sample of limited size. Differences in isokinetic strength parameters between groups will be analyzed using one-way analysis of variance or non-parametric equivalents when appropriate. Associations between Wingate-derived anaerobic parameters and isokinetic strength measures will also be examined using correlation analyses.

The results of this study are expected to clarify whether individuals with higher anaerobic power levels demonstrate superior isokinetic knee extensor and flexor strength profiles. The findings may contribute to a better understanding of the interaction between anaerobic performance capacity and lower-extremity muscle strength, with potential implications for performance profiling, training program design, and exercise-based rehabilitation strategies in recreationally active populations.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged between 20 and 30 years

  * Moderately physically active individuals, as defined by the International Physical Activity Questionnaire (IPAQ)
  * Apparently healthy, with no known neurological, vestibular, or musculoskeletal disorders affecting balance
  * Ability to stand independently and complete balance assessments
  * Willingness to participate and provide written informed consent

Exclusion Criteria:

* History of lower-limb, spine, or pelvic injury or surgery within the past 6 months

  * Presence of acute or chronic pain affecting posture or balance
  * Diagnosed neurological, vestibular, or balance disorders
  * Use of medications or substances that may affect neuromuscular function or postural control
  * Participation in another clinical or observational study within the past 3 months

Ages: 20 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of recreationally active young adult males aged 22-30 years who engage in regular physical activity at least two days per week. Participants will be non-elite individuals without a history of serious orthopedic injury within the past six months, cardiovascular or respiratory disease, or regular medication use. All participants will be healthy volunteers capable of performing maximal exercise testing and will provide written informed consent prior to participation.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic knee extensor and flexor peak torque (Nm) at 60°/s | day 1 (Assessed during a single laboratory testing session.)
  Peak torque values of the knee extensor and flexor muscles will be assessed using isokinetic dynamometry during concentric contractions at an angular velocity of 60°/s. Measurements will be obtained from the dominant leg following a standardized warm-up protocol. Peak torque (Nm) will be used as the primary indicator of maximal dynamic muscle strength.

SECONDARY OUTCOMES:
Wingate-derived anaerobic performance parameters | day 1 (Assessed during a single laboratory testing session.)
  Anaerobic performance will be assessed using the 30-second Wingate Anaerobic Test performed on a cycle ergometer. Relative peak power (W/kg) will be used.

IPD SHARING:
Plan to Share IPD: No
This observational study will follow a cross-sectional group comparison design. Eligible participants will undergo body composition assessment, isokinetic knee extensor and flexor strength testing, and a 30-second Wingate Anaerobic Test conducted on separate days. Based on relative peak power (W/kg) derived from the Wingate test, participants will be classified into low, moderate, and high anaerobic power groups. Isokinetic strength parameters will be compared across groups, and associations between anaerobic performance and muscle strength measures will be analyzed to address the study objectives.

REFERENCES:
- [Background] Bar-Or O. The Wingate anaerobic test. An update on methodology, reliability and validity. Sports Med. 1987 Nov-Dec;4(6):381-94. doi: 10.2165/00007256-198704060-00001. No abstract available. PMID 3324256
- [Background] Zupan MF, Arata AW, Dawson LH, Wile AL, Payn TL, Hannon ME. Wingate Anaerobic Test peak power and anaerobic capacity classifications for men and women intercollegiate athletes. J Strength Cond Res. 2009 Dec;23(9):2598-604. doi: 10.1519/JSC.0b013e3181b1b21b. PMID 19910814
- [Background] Park JH, Kim JE, Yoo JI, Kim YP, Kim EH, Seo TB. Comparison of maximum muscle strength and isokinetic knee and core muscle functions according to pedaling power difference of racing cyclist candidates. J Exerc Rehabil. 2019 Jun 30;15(3):401-406. doi: 10.12965/jer.1938180.090. eCollection 2019 Jun. PMID 31316932
- [Background] 1.Alemdaroğlu, U. (2012). The Relationship Between Muscle Strength, Anaerobic Performance, Sprinting Ability, Agility and Vertical Jump Performance. Journal of Strength and Conditioning Research. 2. Bar Or, O. (1987). The Wingate anaerobic test: an update on methodology, reliability, and validity. Sports Medicine, 4(6), 381-394. (aracı olarak anılmış çalışmalarda referans). 3. Castaneda, A., Inbar, O., Bar Or, O. vd. (2021). The Wingate Anaerobic Test: A Narrative Review of the Protocol Variables that Affect the Results Obtained. Applied Sciences, 11(16), 7417. 4. Comin, A. C., vd. (2011). Validity of the Wingate Anaerobic Test for the Evaluation of Anaerobic Power and Capacity. Journal of Strength & Conditioning Research. (Özet referans) 5. Evans, E. M., & Quinney, H. A. (2003). Wingate Anaerobic Test peak power and anaerobic capacity classification system in NCAA athletes. Journal of Strength and Conditioning Research. 6. Harbili, S. (2015). Relationship between lower extremity isokinetic strength and anaerobic power in weightlifters, basketball and soccer players. International Education Studies. 7. Harbili, S. (2022). Comparison of bilateral isokinetic and isometric strength of knee extensor and flexor muscles. European Journal of Exercise & Rehabilitation. 8. Kin İsler, A., vd. (2008). The relationship between anaerobic performance, muscle strength and sprinting ability. International Education Studies. 9. Kavaliauskas, M., & Phillips, S. M. (2016). Reliability and sensitivity of the 6 and 30 second Wingate tests in physically active males and females. Isokinetics and Exercise Science, 24(4), 277-284. 10. Park, J., vd. (2019). Comparison of maximum muscle strength and isokinetic muscle functions according to pedaling power. PMC. 11. Zagatto, A. M., Beck, W. R., & Gobatto, C. A. (2009). Validity of the Running Anaerobic Sprint Test (RAST) for assessing anaerobic power and predicting short-distance performances. Journal of Strength and Conditioning Research, 23(6), 1820-1827. https://doi.org/10.1519/JSC.0b013e3181b3df32 12. Lehance, C., et al. (2009). Muscular strength, functional performances and injury risk in soccer players. Scandinavian Journal of Medicine & Science in Sports. 13. Castaneda, A., vd. (2021). The Wingate Anaerobic Test: A Narrative Review.